CLINICAL TRIAL: NCT00942734
Title: Phase II Clinical Trial of the Combination of RAD001 and Erlotinib in Patients With Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Trial of RAD001 and Erlotinib With Recurrent Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0567; NCI-2012-01643 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Head And Neck Cancer
Keywords: Head and Neck; Squamous Cell Carcinoma; RAD001; Erlotinib; Everolimus; OSI-774; Tarceva
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 + Erlotinib (Experimental): RAD001 1 tablet (5 mg) by mouth every day of each 28 day study cycle. Erlotinib one tablet (150 mg) by mouth every day of each 28 day study cycle.
  Interventions: Drug: Erlotinib; Drug: RAD001

INTERVENTIONS:
Drug: Erlotinib — One tablet (150 mg) by mouth every day of each 28 day study cycle.
  Other Names: OSI-774; Tarceva
Drug: RAD001 — 1 tablet (5 mg) by mouth every day of each 28 day study cycle.
  Other Names: Everolimus

SUMMARY:
The goal of this clinical research study is to learn if RAD001 in combination with Tarceva (erlotinib hydrochloride) can help to control head and neck squamous cell cancer (HNSCC). The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

RAD001 is designed to stop cancer cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, and this may cause the tumor cells to die.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 1 RAD001 tablet and 1 erlotinib hydrochloride tablet every day of each 28 day study "cycle".

Both drugs should be taken at the same time, by mouth, with a cup (8 ounces) of water. You should take the drugs at least 1 hour before or 2 hours after eating. You should take the study drugs at around the same time each day. Your eating habits around the time you take the drugs should stay the same while you are on study. lf you vomit, you should not take another tablet until your next scheduled dose.

Tell your doctor if you have any side effects, as your dose(s) of study drug(s) may be lowered or stopped for a few days. You may be given drugs to help reduce the risk of side effects.

Study Visits:

On Day 1 (+/- 3 days) of each cycle, the following tests and procedures will be performed:

* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests. If your doctor thinks it is needed, you may have to have these blood tests more often.

On Day 1 (+/- 3 days) of every evenly numbered cycle (Cycles 2, 4, 6, and so on), you will have a CT scan or MRI scan to check the status of the disease.

Length of Study:

You may continue to take the study drugs for as long as you are benefitting. You will be taken off study if the disease gets worse or if you have intolerable side effects.

End-of-Study Visit:

When you go off study for any reason, you will have an end-of-study visit. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a CT scan or MRI scan to check the status of the disease.

Follow-Up:

You will be called within 30 days after the end-of-study visit and asked how you are doing and about any possible side effects that you may have had. The call should take about 5 minutes.

This is an investigational study. RAD001 is FDA approved and commercially available for the treatment of certain types of breast cancer. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of advanced non-small cell lung carcinoma (NSCLC) and advanced pancreatic cancer. The use of this drug combination for the treatment of HNSCC is investigational.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma of the head and neck
2. Patients that have failed one platinum-containing chemotherapy regimen with or without EGFR inhibitor and/or epidermal growth factor receptor (EGFR) inhibitor as systemic therapy for recurrent/metastatic disease. Prior investigational therapy (with the exclusion of mammilian target of rapamycin (mTOR) inhibitor) allowed but at least 4 weeks must have elapsed with recovery from all toxicities
3. Patients who had prior induction or concurrent chemotherapy delivered as part of their primary treatment are eligible as long as they have completed primary therapy at least 6 months prior to study entry.
4. Patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
5. Age >/= 18 years
6. Minimum of two weeks since any major surgery or completion of radiation. Note: Patients may have received prior radiation therapy to tumor sites that will not be assessed for response, unless there is evidence of progression.
7. Completion of all prior systemic anticancer therapy for the treatment of recurrent/metastatic disease (adequately recovered from the acute toxicities of any prior therapy) at least 4 weeks prior to study entry
8. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
9. Laboratory Values (within 14 days prior to administration of study drugs): Adequate bone marrow function as shown by: absolute neutrophil count (ANC) >/= 1.5 * 10^9/L, Platelets >/= 100 * 10^9/L, Hgb > 10 g/dL; Adequate liver function as shown by: serum bilirubin </=1.5 * upper limit of normal (ULN), and serum transaminases activity </= 3 * ULN. With the exception of serum transaminases (< 5 * ULN) if the patient has liver metastases
10. Continued from Inclusion # 9: Fasting serum cholesterol </= 300 mg/dL OR </= 7.75 mmol/L AND fasting triglycerides </= 2.5 * ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
11. Signed informed consent

Exclusion Criteria:

1. Prior treatment with any investigational drug within the preceding 4 weeks, concomitant chemotherapy, hormonal therapy, radiotherapy or immunotherapy, or therapy with agents otherwise used in treatment of cancer (for example, methotrexate for rheumatoid arthritis)
2. Chronic treatment with systemic steroids or another immunosuppressive agent. Steroids will not be allowed and should be discontinued 24 hours prior to initiation of treatment on protocol. An exception for replacement steroids prescribed for adrenal insufficiency will be allowed.
3. Patients should not receive immunization with attenuated live vaccines during study period or within one week of study entry
4. Patients with metastatic disease to the brain, unless treated and controlled and the patient is off steroids and/or antiepileptics for at least 3 weeks.
5. Other malignancies within the past 2 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
6. Patients with active skin, mucosa, ocular or gastrointestinal disorders grade > 1
7. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction, </= 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia
8. Continued from Exclusion #7: severely impaired lung function; uncontrolled diabetes as defined by fasting serum glucose >1.5x ULN; any active (acute or chronic) or uncontrolled infection/ disorders.; nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy; liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
9. A known history of HIV or AIDS-related illness or previous seropositivity for the virus
10. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study agents (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
11. Patients with any condition which impairs the ability to swallow study agent intact
12. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin)
13. Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (Women of childbearing potential (WOCP) must have a negative urine or serum pregnancy test within 7 days prior to administration of study drugs). WOCP: A female of child bearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
14. (Continued from Exclusion # 13) Females must either commit to abstinence from heterosexual intercourse or use a barrier method of contraception. Oral, implantable, and injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Males must either commit to abstinence from heterosexual intercourse or use a barrier method of contraception.
15. Lack of resolution of all toxic manifestations of prior chemotherapy biologic therapy or radiation therapy.
16. Patients who have received prior treatment with an mTor inhibitor.
17. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
18. Patients with psychiatric illness or confusional status that may impair the patient's understanding of the informed consent
19. Patients unwilling to or unable to comply with the protocol
20. Patients with any condition which impairs the ability to swallow study agent intact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vali Papadimitrakopoulou, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Massarelli E, Lin H, Ginsberg LE, Tran HT, Lee JJ, Canales JR, Williams MD, Blumenschein GR Jr, Lu C, Heymach JV, Kies MS, Papadimitrakopoulou V. Phase II trial of everolimus and erlotinib in patients with platinum-resistant recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2015 Jul;26(7):1476-80. doi: 10.1093/annonc/mdv194. Epub 2015 May 29. PMID 26025965
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 17, 2009 to February 08, 2013. Recruitment was done in various medical clinics in the United States.
Pre-assignment Details: Of the forty-nine participants registered, six participants were ineligible and not treated.
Groups:
- RAD001 + Erlotinib: RAD001 5 mg orally and Erlotinib 150 mg orally every day of each 28 day study cycle.
Period: Overall Study
Arm/Group | RAD001 + Erlotinib
Started | 43
Completed | 35
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 3
Not completed — Disease Progression | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 + Erlotinib
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: 12-Week Progression-Free Survival (PFS)
Description: Tumor assessments performed by Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI) after 4 weeks, 12 weeks, then every 8 weeks thereafter. Participants who received at least one dose of RAD001+erlotinib and who die before 12 weeks, counted as having progressive disease. Response Evaluation Criteria in Solid Tumors (RECIST) defined as Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progression-free survival defined as stable disease or better. Progressive Disease (PD): >20% increase in sum of LD of target lesions, taking as reference smallest sum LD recorded since treatment started or appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum LD since treatment started.
Time Frame: 12 weeks
Population: Eight participants were not evaluable.
Measure: Number; unit: Percentage of Participants
Arm/Group | RAD001 + Erlotinib
Number analyzed (Participants) | 35
Percentage of Participants | 48.57

ADVERSE EVENTS:
Time Frame: Adverse events collected through 12 weeks of treatment (± 3 days).
Arm/Group | RAD001 + Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 + Erlotinib (N=43)
hypercalcaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 + Erlotinib (N=43)
ACNE (Skin and subcutaneous tissue disorders) | 27 (27)
ANOREXIA (Gastrointestinal disorders) | 3 (3)
CHOLESTEROL (Metabolism and nutrition disorders) | 2 (2)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 5 (5)
DIARRHEA (Gastrointestinal disorders) | 18 (18)
DIZZINESS (General disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EDEMA: HEAD AND NECK (General disorders) | 9 (9)
EDEMA: LIMB (General disorders) | 2 (2)
FATIGUE (General disorders) | 18 (18)
FEVER WITHOUT NEUTROPINIA (Investigations) | 2 (2)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2)
HEMOGLOBIN (Blood and lymphatic system disorders) | 5 (5)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
LEUKOCYTES (Blood and lymphatic system disorders) | 2 (2)
MUCOSITIS (Gastrointestinal disorders) | 18 (18)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 9 (9)
PAIN (ORAL CAVITY) (Gastrointestinal disorders) | 2 (2)
PLATELETS LEVEL (Blood and lymphatic system disorders) | 5 (5)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (4)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 5 (5)
WEIGHT LOSS (General disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes